CLINICAL TRIAL: NCT03247894
Title: Influence of Obstetric Anesthesia and Analgesia on the Progression of the Disease in Multiple Sclerosis Parturients: Retrospective Cohort Study
Brief Title: Obstetric Anesthesia and Analgesia and Multiple Sclerosis
Acronym: OBAANAMS
Status: Completed | Type: Observational
Sponsor: Brno University Hospital (Other)
Collaborators: Masaryk University (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, doc.MD. Ph.D., Brno University Hospital
Other Study IDs: KDAR FN Brno 2017
Record Dates: First submitted 2017-08-04; First posted 2017-08-14 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis, anesthesia
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MS patients who after labour: Patients with multiple sclerosis after labour in tertiary center was screened for progression of MS in 10 months period after labour
  Interventions: Other: Data search

INTERVENTIONS:
Other: Data search — Patients data were searched for the patients with MS, who laboured in tertiary perinatology center in the study period

SUMMARY:
Aim of the retrospective study was to evaluate the influence of the labour on the clinical course of the parturients with MS in selected 6 month follow-up interval and to evaluate to possible influence of the different anesthesia/analgesia types on the course of MS.

DETAILED DESCRIPTION:
The role of anesthesia in multiple sclerosis (MS) progression remains unclear in spite of few foreign studies. The most frequently afflicted patients by MS are women of childbearing age and influence of anesthesia or obstetric epidural analgesia has only not been investigated in Czech Republic. The study aims to retrospectively compare the further course of the disease of MS in patients who labor between 2004 and 2013 in University Hospital Brno either by caesarean section or vaginally with epidural analgesia , with patients who gave birth spontaneously without anesthesia.The aim of the study was to evaluate the influence of the labour on the clinical course of MS and further evaluate the possible influence of the type of anesthesia/analgesia in the peripartal period on the MS progression.

ELIGIBILITY:
Inclusion Criteria:

* Parturients with multiple sclerosis
* Possible follow up - neurologic examination available after 10 month from delivery

Exclusion Criteria:

* probable or no multiple sclerosis at time of labor
* unknown neurology history
* unknown data on neurology outcome 6 months after labour
* Incomplete data
* Follow-up not possible

Ages: 18 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Parturients with multiple sclerosis
Study Population: Parturients with multiple sclerosis after labour in tertiary perinatology center
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Multiple sclerosis decompensation/progression at 3rd month | 3 months after labour
  Relapse occurence from labour to 3 months, after delivery was recorded. A relapse was defined as the appearance or worsening of symptoms of neurologic dysfunction lasting more than 24 hours, new lesions on MRI or need of reinforcement in treatment. For disease state after delivery we used dichotomic approach: relapse (at least one) or no relapses.
Multiple sclerosis decompensation/progression | 3 months after labour
  Relapse occurence from labour to 6 months after delivery

SECONDARY OUTCOMES:
MS progression and the type of anesthetic method | 6 months after labour
  MS progression comparison due to the type of anethesia

CONTACTS AND LOCATIONS:
Locations (1):
- Brno University Hospital, Brno, Czechia, 62500, Czechia, Czechia

IPD SHARING:
Plan to Share IPD: Undecided